CLINICAL TRIAL: NCT00988975
Title: Does Pelvicol Graft in the Posterior Compartment Offer Any Benefit to Surgical Outcomes During Laparoscopic Sacral Colpoperineopexy?
Brief Title: Trial to Determine Which of Two Surgical Techniques Works Better to Correct Vaginal Bulging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Urogynecology Associates, Indiana (Other)
Responsible Party: Douglass Hale, MD, Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-046
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Rectocele
MeSH Terms: conditions — Rectocele

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvicol graft (Active Comparator)
  Interventions: Procedure: Insertion of pelvicol graft
- No graft material (No Intervention): No graft material

INTERVENTIONS:
Procedure: Insertion of pelvicol graft — Pelvicol graft
  Arms: Pelvicol graft

SUMMARY:
Women with vaginal bulging who are undergoing laparoscopic sacrocolpopexy at Clarian Health are eligible to enroll in this study. Two different methods of correcting rectocele at the time of sacrocolpopexy will be compared for surgical outcome, surgical complications, and patient satisfaction with intercourse and bowel function. One of the surgical methods uses an additional graft material and one surgical method does not. It is hypothesized that the method which uses an additional graft material to strengthen the patient's tissues will have a better outcome.

ELIGIBILITY:
Inclusion Criteria:

* women with stage 2 pelvic organ prolapse undergoing laparoscopic sacrocolpopexy

Exclusion Criteria:

* concomitant colo-rectal procedure
* allergy to pork
* any contraindication to laparoscopic sacrocolpopexy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Anatomic success of rectocele repair | 6 months

SECONDARY OUTCOMES:
change in patient symptomatology post-operatively | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clarian North, Carmel, Indiana
  - Clarian Methodist, Indianapolis, Indiana